CLINICAL TRIAL: NCT01875822
Title: Open Label Study of Curcumin C-3 Complex, the Prototypal Epigenetic Modulator, as an Augmentation Strategy to Antipsychotic Therapy,for Improving Negative Symptoms and Cognition in Schizophrenia
Brief Title: Open-label Study of Curcumin C-3 Complex in Schizophrenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Woodbury, Michel, M.D. (Individual)
Collaborators: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06T-773; 719-325-8400 [Coast] (Other: Coast Inc. IRB Board review assigned number)
Record Dates: First submitted 2013-06-04; First posted 2013-06-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Depression
Keywords: Curcumin; Epigenetics; Schizophrenia; Nitric Oxide synthetase; cognition; negative symptoms
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supercurcumin (Experimental): The study protocol stipulates that subjects diagnosed as DSM IV-TR (Diagnostic Statistical Manual IV-Transitional Revised) would be receiving either 1 gm Super-Curcumin@ capsule once daily or 4 gm Super-Curcumin@ once daily for a total of 16 weeks. Super-Curcumin@ in capsule form is a patented formulation of curcumin certified by Sabinsa Corp.NJ USA and produced by America's Finest Inc. 1 gm-capsule Super-Curcumin@ consist of 1 gm Curcumin C-3 complex and 5 mg of Bioperine.
  Interventions: Dietary Supplement: Super-Curcumin

INTERVENTIONS:
Dietary Supplement: Super-Curcumin — The investigators are comparing the effects of the two dosages of Super-Curcumin@ capsules in the sample of subjects diagnosed as DSM IV-R schizophrenia
  Other Names: Super-Curcumin@: Curcumin C-3 complex and Bioperine

SUMMARY:
Current evidence suggests that schizophrenia as a serious and complex psychiatric disorder, continues to challenge mental health professionals in their search for better treatment options in the community. In the present study, the investigators hypothesized that in patients diagnosed as schizophrenia, adjunct treatment with Curry extract from the plant labeled by botanists as Curcuma Longata, formulated as Super-Curcumin@ , would bring about :1)positive behavioral changes in areas of socialization, emotional well-being, verbal communication and motivation; 2)improvement in measures of memory. Throughout the study, the proprietary product, Super-Curcumin@ consisting of Curcumin C-3 complex combined with the black pepper extract Bioperine to boost the effects of Curcumin. The study was developed to examine whether Curcumin's interaction with the two major signal pathways in the brain regulating brain-behavior: the epigenetic signal (histone modification) and the anti-inflammatory signal (inducible nitric oxide synthetase)in preclinical models is translated to beneficial effects in the treatment of schizophrenia.

DETAILED DESCRIPTION:
Detailed Description: The overall objective of the study was to evaluate whether the standardized proprietary formulation of curcumin [Super Curcumin@ :C-3 Complex@ with Bioperine@) manufactured by American Finest Inc. NJ USA ] extracted from the curry plant (Curcuma Longata) , can improve the negative symptoms and cognitive impairments in patients diagnosed as schizophrenia and to determine the response rate in negative symptoms at 16 weeks. Response rate was defined as the positive change of minimum 30% or higher from baseline to the score measured at 16 weeks. Negative symptoms refer to the cluster of symptoms of apathy, alogia, blunted affect and lack of motivation affecting severely the ways the individual functions in the community at large. In the study, the investigators proposed to test the hypothesize that Super curcumin@ is efficacious and safe when combined with standard antipsychotic drugs in the cohort of patients diagnosed as schizophrenia. Throughout the study, the proprietary product(Super curcumin@) was used. Supercurcumin@ consisted of the primary medicinally active ingredient, Curcumin C-3 Complex, in combination with Bioperine@, the metabolic enhancer extracted from black pepper, in order to increase the systemic bioavailability of curcumin C-3 complex. For the oral formulation of Super- curcumin@: 1 gm-capsule has 1 gm of curcumin C-3 complex and 5 mg of Bioperine@ . The study protocol consisted of recruiting subjects with diagnosed as schizophrenia who would be receiving either 1 gm or 4 gm of Super-Curcumin@ given orally once daily for 16 weeks, on negative symptoms and cognition. For assessing the safety and tolerability of Supercurcumin@ , the study protocol required that the patients would be monitored regularly for vital signs:blood pressure, pulse,body weight, routine blood chemistry and comprehensive adverse events profile (Treatment Emergent Adverse Events checklist) including the AIMS (Abnormal Involuntary Movement Scale). At baseline and at regular intervals throughout the 16-week treatment period, standardized measures of negative and positive symptoms and neurocognition would be administered to examine the efficacy of Curcumin C-3 complex in schizophrenia. For analysing the results, within-subject pre- and post-treatment responses would be subject to statistical procedures to evaluate whether Super-Curcumin@ can ameliorate the persistent negative symptoms and cognitive deficits in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female:
* DSMIV (Diagnostic Statistical Manual -TR version) Schizophrenia
* Male or Female ,
* age 18-65 yrs
* SANS (Scale of Negative Symptoms of Schizophrenia ) > 30
* Stable antipsychotic dosage at least 1 month

Exclusion Criteria:

* Current Substance use Disorder except Nicotine dependence
* Regular Use of NSAID (non-steroidal anti-inflammatory drugs)
* cancer History
* Recent myocardial infarction
* Unstable angina,
* untreated or severe hypertension
* Poorly controlled diabetes mellitus Type I or Type II
* Chronic liver & gallbladder diseases
* Recent GERD (Gastroesophageal Reflux Disorder)
* Pregnancy and breast-fed.
* Allergic reaction to Curcumin
* Neurological disorders: epilepsy, stroke
* Hamilton Depression Scale Hamilton Depression Rating Scale( HAM-D-17 item) > 24 -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Negative Symptoms | Change from baseline Negative symptom at 16 weeks
  PANSS (Positive and Negative Symptom scale).
  The PANSS has three subscales:
  1.Positive symptoms Subscale: delusions, hallucinations , and bizarre behavior; 2.Negative symptoms Subscale: alogia, anhedonia, social withdrawal, lack of motivation 3.General psychopathology Subscale: social interactions, anxiety, sleep, energy level
  --------------------------------------------------------------------------------

SECONDARY OUTCOMES:
Neurocognition measures | Change from Baseline neurocognitive measures at 16 weeks
  The CNS Vital Sign@ is a standardized computerized battery of neurocognitive tests to be administered by trained research personnel to measure neurocognitive domains of memory, attention, logical reasoning, visual-spatial function and executive function.
Positive symptoms | Change from Basline Positive symptoms at 16 weeks
  PANSS (Positive subscale) to measure the positive symptoms: hallucinations, delusions, bizzare behavior and disorganized thoughts
General psychopathology | Change from baseline general psychopathology at 16 weeks
  The BPRS is a standardized psychiatric rating scales to measure symptoms of general psychopathology, depression, anxiety, psychosis and somatic symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Woodbury Farina, MD ABPN, Study Director — University Puerto Rico San Juan PR (US)
Locations (1):
- Dr. Michel Woodbury-Farina, San Juan, Puerto Rico